CLINICAL TRIAL: NCT02476461
Title: Prospektiv Randomisert Sammenlikning Mellom Percutan nålefasciotomi og Xiapex for Dupuytrens Kontraktur
Brief Title: Prospective Randomized Trial Between Needle Fasciotomy and Xiapex for Dupuytrens Contracture
Acronym: PNFvsxiapex
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1234
Record Dates: First submitted 2015-06-05; First posted 2015-06-19 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-04

CONDITIONS: Dupuytrens Contracture
Keywords: percutanepus needle fasciotomy; xiapex; clostridium histolyticum
MeSH Terms: conditions — Dupuytren Contracture | interventions — xiapex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- xiapex (Active Comparator): 1: xiapex: 0,58 mg clostridium histolyticum administered in the dupuytrens cord as discribed in producers manual
  Interventions: Drug: xiapex
- PNF (Experimental): percutaneous needle fasciotomi is performed at affected cords
  Interventions: Procedure: percutaneous needle fasciotomy

INTERVENTIONS:
Drug: xiapex
  Other Names: clostridium histolyticum
  Arms: xiapex
Procedure: percutaneous needle fasciotomy
  Other Names: PNF
  Arms: PNF

SUMMARY:
The purpose of this study is to investigate whether percutaneous needle fasciotomy is as effective for treating Dupuytrens contracture as Xiapex. Immidiate treatment effect is to be investigated, as iskontracture size after 5 years. Contracture size after one and three years, and subjective hand function is also to be investigated.

DETAILED DESCRIPTION:
Prospective randomized study between Percutanous Needle Fasciotomy and Xiapex for Dupuytrens contracture.

A total of 50 patiens are to be randomized to eighter percutaneous needle fasciotomy or Xiapex treatment.

The patients randomized to xiapex treatment are treated as described in the product manual. Extentin treatment after one day.

The patients randomized to percutaneous needle fasciotomy are treated with the cutting teqnique: A littel quaddle local anestesia (xylocaine with adrenaline) is to be injected subcutant over the cord. After thet we use a 19G needle to cut the cord sufficient number sites to extend the finger.

The patients will be follwed up at 3 weeks, 3 months, 1 year, 3 years and 5 years. Investigators record contracture size, quicq-DASH, pain (VAS) and hand disability (VAS) pretreatment and at all controlls. At 3 weeks investigators register procedure complain. Side effects and complications, and advere effects are also to be investigated.

Our hypothesis is that it is no difference between the two methods in regard of contracture size after five years.

Inclution criteria: Symptomatic primary Dupuytrens contracture with palpable cord in one to three fingers, involving MCP, and total contracture size is over 30 degrees. Patient age over 18 years.

Exclution criteria:

Previously treated Dupuytrens contracture in the same hand more than tree affected fingers we will not include thumbs Other symptomatic injury or disease influencingf hand function ASA>3 Expected lifetime less than five years tetracycline treatment within two weeks pregnancy nursing allergy to clostridium histolyticum concmittent other clinical trial

ELIGIBILITY:
Inclusion Criteria:

* symptomatic Dupuytrens contracture with palpable cord, involving MCP, total contracture size over 30 degrees

Exclusion Criteria:

* previous treated dupuytrens contracture same hand
* more than tree fingers involvement
* we will not include thumbs
* other things affecting hand function
* ASA>3
* expected to live under five years
* Tetracycline treatment within two weeks
* pregnancy
* nursing
* allergy to clostridium histolyticum
* participant in other trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
contracture size (degrees) | five years

SECONDARY OUTCOMES:
contracture size | post treatment
  Contracture size mesured in degrees in each finger joint

OTHER OUTCOMES:
contracture size (degrees) | one year
  contracture size mesured in degrees in each finger joint
contracture size (degrees) | three years
  contracture size mesured in degrees in each finger joint
quick-Dash | one, three and five years
  Quick-DASH functional score measured in points.
Pain | one, three, five years
  Visual Analogue score
Hand disability | oen, three, five years
  Visual Analogue score

CONTACTS AND LOCATIONS:
Overall Officials: hallgeir bratberg, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo Universitetssykehus, Oslo, Oslo County, Norway